CLINICAL TRIAL: NCT02797262
Title: Measuring and Monitoring Adherence to ART With Pill Ingestible Sensor System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Yale University (Other); University of Nebraska (Other)
Responsible Party: Principal Investigator, Honghu Liu, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1R01MH110056 (NIH)
Record Dates: First submitted 2016-06-01; First posted 2016-06-13 (Estimated); Results first posted 2021-12-20 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: HIV/AIDS; Medication Adherence
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Medication Adherence | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Intervention (Experimental): Building on the available Proteus devices, the investigators will design and create a Proteus digital health feedback (PDHF) system to transmit the adherence data using mobile technology to allow treatment monitoring that is, direct confirmation of the type, dose, date and time of oral pharmaceutical ingestion using wirelessly observed therapy (WOT).
  The investigators will test overall utility (including feasibility, acceptability and sustainability) of the PDHF system, its accuracy for measuring adherence and its impact on enhancing patients' level of adherence and the effect on virologic and clinical outcomes (exploratory), the retention of its impact on keeping up with adherence and improvement of plasma HIV RNA and CD4 cell count after the 16-week usage of the PDHF system.
  Interventions: Device: Proteus digital health feedback (PDHF) system
- Control (No Intervention): UC is chosen as the control condition because it meets ethical and moral requirements to attempt treatment. Eligible patients will be randomized to one of the two conditions using a stratified urn randomization procedure to increase the likelihood of balanced allocation of prognostic variables at baseline.

INTERVENTIONS:
Device: Proteus digital health feedback (PDHF) system — Building on the available Proteus devices, the investigators will design and create a PDHF system to transmit the adherence data using mobile technology to allow treatment monitoring that is, direct confirmation of the type, dose, date and time of oral pharmaceutical ingestion using wirelessly observed therapy (WOT).
  Arms: Intervention

SUMMARY:
Introduction of antiretroviral therapy (ART) has transformed HIV-infection from a fatal to manageable disease but adherence to ART remains critical to optimize outcomes. Existing measures of ART adherence provide only inferred measures of actual drug intake and most offer no real-time notification capability. Directly observed therapy measures actual drug intake but is not practical. These limitations constrain research into medication adherence and more importantly, limit our ability to develop real-time interventions based on feasible, in vivo monitoring of adherence among HIV-infected people to facilitate medication-taking. The Proteus digital health feedback (PDHF) system, a pill ingestible sensor based adherence measuring and monitoring system developed by Proteus Digital Health, addresses these limitations. It involves use of an ingestible sensor, a tiny edible material that is over-encapsulated along with prescribed medication. The sensor is activated by ingestion and is sensed by a patch worn by the patient with an embedded monitor and sensor. The monitor sends a Bluetooth signal to a mobile device, which in turn sends an encrypted message to a central server, thus effecting real-time monitoring that a dose has been taken. The investigators propose to develop a data receiving hub and add to these components an automated text message that is sent to the patient when a dose is missed. The investigators will evaluate the feasibility, acceptability and sustainability of using the PDHF system; assess the accuracy of the PDHF system in measuring adherence to ART; and evaluate the efficacy of the PDHF system for monitoring and leveraging adherence to ART.

DETAILED DESCRIPTION:
Introduction of antiretroviral therapy (ART) has transformed HIV-infection from a fatal to manageable disease but adherence to ART remains critical to optimize outcomes. Existing measures of ART adherence such as self-report, pill counts, electronic pill-bottle caps, and prescription refills, provide only inferred measures of actual drug intake and most offer no real-time notification capability. Directly observed therapy measures actual drug intake but is not practical. These limitations constrain research into medication adherence and more importantly, limit our ability to develop real-time interventions based on feasible, in vivo monitoring of adherence among HIV-infected people to facilitate medication-taking. The Proteus digital health feedback (PDHF) system, a pill ingestible sensor based adherence measuring and monitoring system developed by Proteus Digital Health, addresses these limitations. It involves use of an ingestible sensor, a tiny edible material that is over-encapsulated along with prescribed medication. The sensor is activated by ingestion and is sensed by a patch worn by the patient with an embedded monitor and sensor. The monitor sends a Bluetooth signal to a mobile device, which in turn sends an encrypted message to a central server, thus effecting real-time monitoring that a dose has been taken. The investigators propose to develop a data receiving hub and add to these components an automated text message that is sent to the patient when a dose is missed. The ingestible sensor and patch monitor system is already FDA-approved as safe, but has yet to be tested in HIV-infected patients in clinical setting. The first goals of this study are to confirm the bioavailability of over-encapsulated antiretrovirals (ARVs) and to pilot-test the use of the PDHF system in 15 participants prescribed ARVs to test and identify approaches that optimize the use of this measuring and monitoring system. The next goals are to determine the system's feasibility, acceptability, sustainability, accuracy and efficacy in fostering ART adherence. Feasibility, acceptability and sustainability will be assessed by patients' rating of the system and the rate of dropping off from using the system. Accuracy will be evaluated by the associations between adherence to ART measured by the PDHF system and other adherence measures such as plasma drug level concentrations of ARVs and self-report. Efficacy will be assessed by comparing adherence of participants assigned to the PDHF system and participants assigned to usual care (UC) over time, with exploratory outcomes of viral load and cluster of differentiation 4 (CD4). The investigators will recruit 120 of HIV-infected patients 18 years or older with sub-optimal adherence. Participants will be randomized to receive the PDHF system or UC for 16 weeks with monthly assessments. The durability of effects of the PDHF system after stopping the use of the system will be determined during a 12-week follow-up stage. In summary, The investigators will evaluate the feasibility, acceptability and sustainability of using the PDHF system; assess the accuracy of the PDHF system in measuring adherence to ART; and evaluate the efficacy of the PDHF system for monitoring and leveraging adherence to ART.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected individuals in HIV care
* greater than 17 years of age
* demonstrated ability to take over-encapsulated ARVs at time of screening; able to provide informed consent
* On ART with sub-optimal adherence estimated by either patient (self-reports < 90% adherence over last 28 days) or treating clinician (e.g., based on gaps in treatment (e.g., missed appointments) or viral load elevations within last 6 months)

Exclusion Criteria:

* Inability to follow the study procedures manifested during the intake, as evidenced by mental confusion, disorganization, intoxication, withdrawal, risky or threatening behavior

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Honghu Liu, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- LA BioMed, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available within 6 months of study completion.

REFERENCES:
- [Derived] Wang Y, Daar ES, Huang Y, Xiong D, Shen J, Zhou L, Siqueiros L, Guerrero M, Rosen MI, Liu H. Adherence to Antiretrovirals and HIV Viral Suppression Under COVID-19 Pandemic Interruption - Findings from a Randomized Clinical Trial Using Ingestible Sensors to Monitor Adherence. AIDS Behav. 2023 Dec;27(12):4041-4051. doi: 10.1007/s10461-023-04118-9. Epub 2023 Jul 4. PMID 37401993

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Building on the available Proteus devices, the investigators will design and create a Proteus digital health feedback (PDHF) system to transmit the adherence data using mobile technology to allow treatment monitoring that is, direct confirmation of the type, dose, date and time of oral pharmaceutical ingestion using wirelessly observed therapy (WOT).
  The investigators will test overall utility (including feasibility, acceptability and sustainability) of the PDHF system, its accuracy for measuring adherence and its impact on enhancing patients' level of adherence and the effect on virologic and clinical outcomes (exploratory), the retention of its impact on keeping up with adherence and improvement of plasma HIV RNA and CD4 cell count after the 16-week usage of the PDHF system.
  Proteus digital health feedback (PDHF) system: Building on the available Proteus devices, the investigators will design and create a PDHF system to transmit the adherence data using mobile technology to allow treatment monitoring that is, direct confirmation of the type, dose, date and time of oral pharmaceutical ingestion using wirelessly observed therapy (WOT).
- Control: Usual care (UC) is chosen as the control condition because it meets ethical and moral requirements to attempt treatment. Eligible patients will be randomized to one of the two conditions using a stratified urn randomization procedure to increase the likelihood of balanced allocation of prognostic variables at baseline.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 65 | 65
Baseline | 54 | 58
Completed | 45 | 54
Not Completed | 20 | 11
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Lost to Follow-up | 10 | 7
Not completed — Death | 1 | 2
Not completed — Adverse Event | 1 | 0
Not completed — COVID-19 | 2 | 1
Not completed — Out-of-country | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 54 | 58 | 112
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 53 | 54 | 107
  >=65 years | 1 | 4 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (11.1) | 45.7 (12.4) | 46.2 (11.8)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 5 | 5 | 10
  Gender: Male | 44 | 43 | 87
  Gender: Transgender: Male to Female | 5 | 10 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race and Ethnicity: White | 6 | 8 | 14
  Race and Ethnicity: Black | 24 | 30 | 54
  Race and Ethnicity: Latino | 19 | 16 | 35
  Race and Ethnicity: Asian | 1 | 1 | 2
  Race and Ethnicity: Other | 4 | 3 | 7
Education [Count of Participants; unit: Participants]
  8th grade or less/ Some high school but did not graduate | 8 | 10 | 18
  High school graduate/ Some college but no degree | 38 | 39 | 77
  Completed college/ More than four-year college degree | 8 | 9 | 17
Employment [Count of Participants; unit: Participants]
  Part-time/full-time | 9 | 19 | 28
  None/full-time student/retired/disabled | 45 | 39 | 84
HIV+ Years [Mean (Standard Deviation); unit: years] | 14.5 (8.0) | 14.0 (9.3) | 14.2 (8.7)
Years under Antiretroviral Treatment [Mean (Standard Deviation); unit: years] | 12.6 (7.5) | 11.6 (7.7) | 12.0 (7.6)
History of AIDS Diagnosis [Count of Participants; unit: Participants]
  Yes | 12 | 12 | 24
  No | 42 | 46 | 88
Detectable Viral Load at Baseline [Count of Participants; unit: Participants]
  Less than 50 copies/mL | 35 | 46 | 81
  Greater than 50 copies/mL | 19 | 12 | 31

OUTCOME MEASURES:

1. Primary Outcome: Adherence Measured by Sensor by Percentage of Prescribed Medications Taken
Description: Adherence to antiretroviral therapy (ART) measured by Proteus digital health feedback (PDHF) system for 16 weeks, including percent of prescribed medication taken.
Time Frame: Adherence to ART measured by PDHF system for 16 weeks
Measure: Mean (Standard Deviation); unit: percentage of prescribed medication
Arm/Group | Intervention
Number analyzed (Participants) | 54
percentage of prescribed medication | 87.5 (33.1)

2. Primary Outcome: Pharmacokinetic Adherence by Integrated Pharmacokinetic Adherence Score
Description: The plasma concentration-time data of tenofovir (TFV) from participants who have a tenofovir alafenamide (TAF) in their regimen are used to quantify intra-patient pharmacokinetic (PK) variability as a measure of adherence. Plasma concentrations of TFV are measured by liquid chromatography/tandem mass spectrometry. A population PK model will be developed using a nonlinear mixed-effects approach with data from all the time points. The integrated PK adherence score (IPAM) will be calculated. The IPAM score ranges from 0 to 1. A high score indicates high concentration predictability and relatively higher adherence, while a low score indicates low predictability and lower adherence.
Time Frame: Blood samples will be obtained in all participants before and 2 and 6 hours following an observed dose (baseline) and then at weeks 4, 8, 12, 16, 20, 24 and 28.
Population: For the trial phase, we pick the most common drug with the longest plasma half-life to use for the PK-based method of adherence. That ended up being tenofovir alafenamide (TAF). Only 86 of the participants in the final analysis had available data for the PK analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 44 | 42
score on a scale | 0.817 (0.276) | 0.798 (0.267)
Statistical Analysis 1: Comparison: Intervention vs Control; Compared the IPAM score between two groups; Test type: Superiority; p = 0.57, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p = 0.05; Mean Difference (Net) = 0.02 — Treatment Difference = Intervention - Control

3. Primary Outcome: Self-Reported Medication Adherence and "Change" Over Time
Description: The investigators will use a widely-used measure of self-reported adherence for percent of prescribed dose taken during the preceding seven days. This tool is easy to use and has been significantly associated with virological and immunological outcomes. Due to its potential bias, self-reported adherence will be calibrated by drug level concentration to leverage its accuracy and used in analysis when calibrated self-report adherence is appropriate to be used.
Time Frame: Self-report adherence will be measured at baseline, and weeks 4, 8, 12, 16, 20, 24, and 28.
Population: Lost to follow-up, missed visits, or no self-reported adherence.
Measure: Mean (Standard Deviation); unit: percentage of prescribed medication
Arm/Group | Intervention | Control
Number analyzed (Participants) | 54 | 58
percentage of prescribed medication
  Week 0: number analyzed (Participants) | 54 | 52
  Week 0 | 90.7 (14.5) | 87.4 (13.2)
  Week 4: number analyzed (Participants) | 53 | 50
  Week 4 | 91.1 (15.7) | 87.4 (15.2)
  Week 8: number analyzed (Participants) | 50 | 51
  Week 8 | 90.6 (17.0) | 91.6 (13.5)
  Week 12: number analyzed (Participants) | 44 | 48
  Week 12 | 88.3 (17.0) | 82.1 (24.9)
  Week 16: number analyzed (Participants) | 43 | 45
  Week 16 | 88.7 (17.5) | 91.7 (16.3)
  Week 20: number analyzed (Participants) | 43 | 47
  Week 20 | 90.7 (20.9) | 84.5 (23.2)
  Week 24: number analyzed (Participants) | 44 | 46
  Week 24 | 94.8 (8.8) | 87.3 (22.4)
  Week 28: number analyzed (Participants) | 43 | 49
  Week 28 | 93.0 (11.8) | 90.1 (19.8)

4. Secondary Outcome: Viral Load
Description: Viral Load will be measured at baseline, weeks 4, 8, 12, 16, and 28.
Time Frame: Baseline, weeks 4, 8, 12, 16, and 28.
Population: Lost to follow-up, missed visits, or failed to draw blood viral load.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Intervention | Control
Number analyzed (Participants) | 54 | 58
log10 copies/mL
  Week 0 | 2.273 (1.158) | 2.061 (0.954)
  Week 4: number analyzed (Participants) | 52 | 52
  Week 4 | 1.916 (0.793) | 1.906 (0.516)
  Week 8: number analyzed (Participants) | 47 | 55
  Week 8 | 1.851 (0.680) | 1.916 (0.711)
  Week 12: number analyzed (Participants) | 46 | 50
  Week 12 | 1.873 (0.653) | 1.937 (0.671)
  Week 16: number analyzed (Participants) | 46 | 51
  Week 16 | 1.895 (0.691) | 1.988 (0.895)
  Week 28: number analyzed (Participants) | 42 | 51
  Week 28 | 1.957 (0.816) | 2.230 (1.117)
Statistical Analysis 1: Comparison: Intervention vs Control; Compared the change of the plasma HIV RNA levels during the intervention period (week 0-16) between two groups; Test type: Superiority; p = 0.08, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; Mean Difference (Net) = -0.02 — Treatment Difference = Intervention - Control
Statistical Analysis 2: Comparison: Intervention vs Control; Compared the change of the plasma HIV RNA levels during the post-intervention period (week 16-28) between two groups; Test type: Superiority; p = 0.23, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; Mean Difference (Net) = -0.02 — Treatment Difference = Intervention - Control
Statistical Analysis 3: Comparison: Intervention vs Control; Compared the plasma HIV RNA levels during week 4-28 between two groups; Test type: Superiority; p = 0.03, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; Mean Difference (Net) = -0.73 — Treatment Difference = Intervention - Control

5. Secondary Outcome: Cluster of Differentiation 4 (CD4)
Description: CD4 cell count is a test that measures the number of CD4 cells (a type of the human T-lymphocyte cells) in a HIV patient's blood. The absolute CD4 cell count is measured by a simple blood test, the results of which are reported as the number of CD4 cells per cubic millimeter of blood. HIV-negative people typically have absolute CD4 cell counts between 600 and 1200 cells per cubic millimeter. HIV is a fatal infection, characterized by the targeting and destruction of CD4 cells. People with advanced HIV can have 200 or fewer CD4 cells per cubic millimeter.
Time Frame: on: CD4 will be measured at baseline, weeks 4, 8, 12, 16, and 28.
Population: Lost to follow-up, missed visits, or failed to draw blood CD4.
Measure: Mean (Standard Deviation); unit: cells/cubic millimeters
Arm/Group | Intervention | Control
Number analyzed (Participants) | 54 | 58
cells/cubic millimeters
  Week 0 | 526.17 (279.10) | 542.78 (279.31)
  Week 4: number analyzed (Participants) | 50 | 53
  Week 4 | 531.02 (273.85) | 553.08 (271.42)
  Week 8: number analyzed (Participants) | 44 | 56
  Week 8 | 522.00 (280.32) | 582.25 (293.29)
  Week 12: number analyzed (Participants) | 44 | 50
  Week 12 | 501.20 (251.46) | 577.20 (295.79)
  Week 16: number analyzed (Participants) | 45 | 50
  Week 16 | 522.91 (273.61) | 562.96 (314.09)
  Week 28: number analyzed (Participants) | 40 | 48
  Week 28 | 538.80 (301.42) | 587.69 (318.24)

ADVERSE EVENTS:
Time Frame: 28 weeks
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 1/57 | 1/58
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/58
Other Adverse Events (participants affected / at risk) | 1/57 | 0/58
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (N=57) | Control (N=58)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
This study included a selected group of individuals willing to participate in the trial. Besides, it was designed as a pilot study in a randomized fashion to gather early information regarding this intervention in HIV-infected individuals. As a result, the sample size was relatively small.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-26): https://cdn.clinicaltrials.gov/large-docs/62/NCT02797262/Prot_SAP_000.pdf